CLINICAL TRIAL: NCT04022330
Title: Protective Gr1low Monocytes and Macrophages in Compensated Cardiac Hypertrophy to Limit Decompensation and Heart Damaging
Brief Title: Protective Monocytes and Macrophages to Limit Decompensation and Heart Damaging
Acronym: PROMOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP190224; 2019-A000751-56 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Left Ventricular Hypertrophy; Cardiac macrophages
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Other)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — The blood sampling will be done just before surgery

SUMMARY:
The working hypothesis is that cardiac macrophages specific for the compensated cardiac hypertrophic phase limit the progression toward the decompensated state of heart failure by promoting an inflammatory environment favouring cardiomyocyte survival and preservation of the pump function. The investigators will perform studies in human plasma and monos, cardiac tissues and macrophages to validate this hypothesis.

DETAILED DESCRIPTION:
Left ventricular hypertrophy (LVH) occurs following acute and chronic phases of ischemic heart disease as well as during pressure and/or volume overload (arterial hypertension, valvular heart disease). Persistence of the pathological stimuli, i.e. pressure and/or volume overload, will ultimately lead to the decompensation of cardiac function described as heart failure (HF). HF is worldwide one of the major healthcare concerns both in terms of the loss of human life and economic burden due to the expanding costs of care for patients with this condition (Ambrosy 2014). HF is associated with cardiomyocyte death, exacerbated inflammatory reaction with ensuing fibrosis and alteration of local angiogenesis. A better understanding of the mechanisms involved in the maintenance of the compensated state and in the transition to heart failure will promote the conception of new pharmacological interventions to prevent or even to reverse the transition to heart failure. Based on preclinical studies, the aim of this study is to advance our knowledge of relevant mechanisms involved in this process.

In an experimental setting in mice, the protective role of macrophages presenting an anti-inflammatory polarization in the progression of isuprel-induced left ventricular hypertrophy to irreversible heart failure has been recently demonstrated (Keck et al., submitted). These findings in the experimental model encourage their confirmation in the clinical setting. In the latter case, new therapeutic strategies can be projected to prevent or even to reverse the transition of compensated cardiac hypertrophy to heart failure.

To this purpose, the investigators will study cardiac tissue and blood sample of patients presenting compensated cardiac hypertrophy compared to those with end-stage heart failure.

Patients undergoing aortic valve replacement associated with septal myomectomy for aortic valve stenosis and asymmetric septal hypertrophy as well as patients with hypertrophic obstructive cardiomyopathy (HOCM) undergoing septal myomectomy are included in the group of compensated cardiac hypertrophy. Patients undergoing heart transplantation or implantation of mechanical life supporting system are included in the group of end-stage heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Patients affiliated to a social security regimen
* Informed signed consent

Group 1 : compensated

• Symptomatic patients with severe aortic valve stenosis associated with asymmetric septal hypertrophy or patients with hypertrophic obstructive cardiomyopathy (HOCM), with echocardiographic transvalvular gradient ≥ 40 mmHg associated with echocardiographic septal/posterior wall thickness ≥ 1.3 ejection fraction ≥ 50%, planned for aortic valve replacement with septal myomectomy or septal myomectomy for HOCM

Group 2 : transition • Symptomatic patients with severe aortic valve stenosis associated with asymmetric septal hypertrophy or patients with hypertrophic obstructive cardiomyopathy (HOCM), with echocardiographic transvalvular gradient ≥ 40 mmHg associated with echocardiographic septal/posterior wall thickness ≥ 1.3 ejection fraction < 50%, planned for aortic valve replacement with septal myomectomy or septal myomectomy for HOCM

Group 3 : decompensated

• End-stage heart failure on the waiting list for cardiac transplantation or undergoing ventricular assist device implantation as a bridge to transplantation

Exclusion Criteria:

* Combined aortic valve replacement and coronary artery bypass grafting or mitral/tricuspid surgery
* Emergency operation
* Acute endocarditis
* Patient unable to give his consent
* Patient deprived of freedom or under legal protection (guardianship or curatorship)
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Identification of the complete spectrum of expressed mRNA of cardiac tissue macrophages. | 18 months from start date
  This complete mRNA profile obtained in patients will be compared to the one found in preclinical studies in mice. The genes that are expressed during compensated cardiac hypertrophy in both human and mouse will be sorted out. The expression of the latter genes will be correlated to the cardiac pump function in order to select in the macrophage transcriptome potential markers of compensated cardiac hypertrophy. The presence of these specific macrophage markers will be investigated on frozen cardiac tissue sections by immune-histochemistry and by real time polymerase chain reaction (rtPCR).

SECONDARY OUTCOMES:
Identification of the complete transcriptome (including surface markers) of circulating monocytes from the blood collected for this project | 24 months from start date
  The transcriptome of circulating monocytes will be identified by mRNA sequencing. This complete mRNA profile obtained in patients will be compared to the one found in preclinical studies in mice and the genes that are expressed during compensated cardiac hypertrophy in both human and mouse will be sorted out. The expression of the latter genes will be correlated to the cardiac pump function in order to select in the circulating monocyte transcriptome potential markers of compensated cardiac hypertrophy. The presence of these specific circulating monocyte markers will be investigated by rtPCR.
Determination of the plasmatic factors in correlation with cardiac macrophage that may be specific for the compensated or decompensated state of left ventricular hypertrophy | 24 months from start date
  Assessment of the presence of plasmatic factors: Based on preclinical studies showing circulating plasmatic markers of the compensated cardiac hypertrophic state, the same biomarkers will be assessed in plasma of the patients by ELISA. The concentration of these plasmatic factors will be correlated to the cardiac pump function in order to select potential markers of compensated cardiac hypertrophy.
mRNA of the circulating monocytes | 24 months from start date
  Characterization of mRNA of the circulating monocytes that in correlation with those of cardiac tissue macrophages may be specific for the compensated or decompensated state of left ventricular hypertrophy and thus protective against transition to heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Reza TAVAKOLI, Dr, Principal Investigator — Pitié-Salpêtrière Hospital (AP-HP)
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France